CLINICAL TRIAL: NCT03198624
Title: A Two-part, Single and Multiple Dose, Parallel Group Study to Assess Safety and Pharmacokinetics of Oral HTL0018318 in Healthy Japanese and Caucasian Subjects
Brief Title: Pharmacokinetics of Oral Capsule in Healthy Japanese vs. Caucasian Subjects
Acronym: HTL0018318
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTL0018318-105; 2017-001245-27 (EudraCT Number); C17011 (Other: Richmond Pharmacology)
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Safety Issues; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part A open label, Part B double blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HTL0018318 Low dose, Part A. (Active Comparator): Part A. 1 single dose on day 1. Discharged on day 4 of Period 1 (following 10 day washout).
  Interventions: Drug: HTL0018318
- HTL0018318 High dose, Part A (Active Comparator): 1 single dose on day 1. Discharged on day 4 of period 2 (following 10 day washout).
  Interventions: Drug: HTL0018318
- HTL0018318 Low dose, Part B (Active Comparator): 1 dose daily for 5 days (5 active doses total). Discharged on day 8 of period 1.
  Interventions: Drug: HTL0018318
- Placebo oral capsule, Part B (Placebo Comparator): 1 dose daily for 5 days (5 active doses total). Discharged on day 8 of period 1.
  Interventions: Drug: Placebo oral capsule
- HTL0018318 High dose, Part B. (Active Comparator): 1 dose daily for 5 days (5 active doses total). Discharged on day 8 of period 2.
  Interventions: Drug: HTL0018318
- Placebo oral capsule, Part B. (Placebo Comparator): 1 dose daily for 5 days (5 active doses total). Discharged on day 8 of period 2.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: HTL0018318 — Part A single dose Part B five doses
  Arms: HTL0018318 High dose, Part A; HTL0018318 High dose, Part B.; HTL0018318 Low dose, Part A.; HTL0018318 Low dose, Part B
Drug: Placebo oral capsule — Part B only
  Other Names: placebo, placebo - cap
  Arms: Placebo oral capsule, Part B; Placebo oral capsule, Part B.

SUMMARY:
This is a single and multiple dose, parallel group study to assess safety and pharmacokinetics of oral HTL0018318 in healthy Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
This is a single and multiple dose, parallel group study to assess safety and pharmacokinetics of oral HTL0018318 in healthy Japanese and Caucasian subjects. The study will be conducted in two parts: (A) single doses of HTL0018318 in healthy, adult, male Caucasian and Japanese subjects; (B) multiple doses of HTL0018318 in healthy, adult, male Caucasian and Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, either Caucasian or Japanese aged ≥20 and ≤40 years.
2. Japanese subjects must have lived outside of Japan for ≤ 5 years in total and be first generation Japanese, defined as born in Japan and having 4 biologic grandparents who are ethnic Japanese.
3. The Caucasian subjects should be distinguished especially by very light to brown skin pigmentation and straight to wavy or curly hair, and should be indigenous to Europe, northern Africa and western Asia. Therefore, the study may include Caucasian subjects from North America, New Zealand, Australia and South Africa.
4. Subjects must have a body mass index (BMI) between 18.0-25.0 kg/m² inclusive.
5. Male subjects, if heterosexually active and with a female partner of childbearing potential or a pregnant or breastfeeding partner, must agree to use barrier contraception (male condom) for the treatment period and for at least 3 months after the end of the systemic exposure of the study drug.
6. Satisfactory medical assessment with no clinically significant or relevant abnormalities.
7. Able to perform spirometry/peak flow with a satisfactory technique at screening.
8. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the International Council of Harmonization Good Clinical Practice (GCP) Guideline E6.
9. An understanding, ability, and willingness to fully comply with study procedures and restrictions

Exclusion Criteria:

1. Any history of any condition associated with cognitive impairment, including but not limited to schizophrenia and dementia.
2. History of epilepsy or seizures of any kind at any time.
3. Current or relevant history of any physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
4. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.
5. Presence or history of drug or alcohol abuse in the last 5 years, or the inability to refrain from alcohol use from 48 hours before screening, dosing and each scheduled visit until the end of the study.
6. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within 3 months prior to the planned first day of dosing.
7. Use of prescription medications within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period, or any over-the-counter (OTC) medication (including multivitamin, herbal, or homeopathic preparations, excluding hormonal contraception, hormone-replacement therapy, and/or an occasional dose of acetaminophen) within 7 days prior to Day 1 of the dosing period.
8. History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
9. Has donated or lost 400 mL blood or more within the last 16 weeks preceding the first day of dosing.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Baseline to 72 hours
  Comparison of pharmacokinetics in plasma
Tmax | Baseline to 72 hours
  Comparison of pharmacokinetics in plasma
Area under the curve | Baseline to 72 hours
  Comparison of pharmacokinetics in plasma

SECONDARY OUTCOMES:
Delay in absorption (Tlag) | Baseline to 72 hours
  Pharmacokinetics in plasma
Rate of elimination | Baseline to 72 hours
  Pharmacokinetics in plasma
Half life (t1/2) | Baseline to 72 hours
  Pharmacokinetics in plasma
Amount excreted in urine | Baseline to 72 hours
  Pharmacokinetics in urine
Fraction of dose eliminated unchanged in urine (fe/F) | Baseline to 72 hours
  Pharmacokinetics in urine
Treatment emergent adverse events (TEAEs) | Up to 14 day post dose
  Safety and tolerability
Number of participants with abnormal physical exam results | Up to 14 day post dose
  Safety and tolerability
Heart Rate | Up to 14 day post dose
  Safety and tolerability
Number of participants with abnormal laboratory values | Up to 14 day post dose
  Safety and tolerability
ECG | Up to 14 day post dose
  Safety and tolerability
Blood pressure | Up to 14 day post dose
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD FFPM, Principal Investigator — Richmond Pharmacology
Locations (1):
- Richmond Pharmacology, London, London Bridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No